CLINICAL TRIAL: NCT06487533
Title: Sensing Physiological Symptoms of Opioid Withdrawal and Cravings in Patients With Opioid Use Disorder
Status: Recruiting | Type: Observational
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Battelle Memorial Institute (Other); Hazelden Betty Ford Foundation (Unknown); National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); The HEAL Initiative (Unknown)
Responsible Party: Sponsor
Other Study IDs: SBM-OWP-09; 1R43DA059448 (NIH)
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Opioid Withdrawal; Opioid Use Disorder
Keywords: Physiological Signals; Opioid; Detoxification; Cravings; Autonomic Nervous System
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples will also be collected for drug screens. Biomarkers collected will include cortisol, melatonin, interleukin-6 (IL-6), and Tumor Necrosis Factor alpha (TNF-α levels).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Opioid Use Disorder: Participants with a history of dependence on prescription or non-prescription opioids
  Interventions: Device: EmbracePlus Smartwatch; Device: Corti Sensor

INTERVENTIONS:
Device: EmbracePlus Smartwatch — The EmbracePlus is worn on the user's wrist and continuously collects raw data via specific sensors. These data can be wirelessly transmitted to a paired mobile device. The data received are analyzed by EmpaDSP, which computes the user physiological parameters. The Care App is responsible for transmitting raw data, device information, Care App-specific information, and computed physiological parameters to the Empatica Cloud. The device supports continuous data collection for monitoring of the following physiological parameters:
  * Peripheral skin temperature
  * Electrodermal activity
  * Blood Oxygen Saturation under no motion conditions
  * Activity associated with movement during sleep.
  The EmbracePlus Watch has been used in previous human subject research studies for bio-physiological data collection in other medical conditions and have confirmed that there is minimal risk to participants. This device is therefore exempt from any IDE requirements.
Device: Corti Sensor — The Corti Wearable is a sweat sensor that is worn continuously measure cortisol, melatonin, tumor necrosis alpha interleukin-6 (IL-6) in the protein analytes in the sweat of participants via electrochemical impedance spectroscopy. The Corti Wearable comprises a plastic reader and a replaceable polymer sweat-sensing strip with zinc oxide (ZnO) coated electrodes that is worn on the participant's forearm. It is manufactured through a screen-printing technique that allows for an affinity-based interaction between a capture probe antibody and the target molecule generating electrochemical activity.
  The Cort Wearable has been used in previous human subject research studies for bio-physiological data collection in other medical conditions and have confirmed that there is minimal risk to participants. This device is therefore exempt from any IDE requirements.

SUMMARY:
The primary objective of this trial is to measure changes in physiologic signals to quantify the status of the autonomic nervous system during opioid withdrawal and cravings.

DETAILED DESCRIPTION:
This is a prospective observational clinical trial in which 20 participants with a history of dependence on prescription or non-prescription opioids will be recruited for collection of physiologic data via wearable sensors during a 14-day inpatient detoxification treatment. The EmbracePlus Smartwatch and Corti Sensor will be worn continuously throughout the 14-day treatment course to detect heart rate, heart rate variability, skin conductance, skin temperature, motion, and cortisol levels.

ELIGIBILITY:
Inclusion Criteria

1. Participant has a recent history of opioid dependence; prescription or non-prescription
2. Participant is currently taking, or plans to initiate, medications for opioid use disorder (MOUD)
3. Participant is between 18 and 50 years of age
4. Participant is English proficient
5. Participant is able to provide informed consent and function at an intellectual level sufficient for study requirements
6. Participant is willing to wear wearable sensors for 14 days

Exclusion Criteria

1. Participant presents current evidence of an uncontrolled and/or clinically significant medical condition or psychiatric condition
2. Participant has a history of epileptic seizures
3. Participant has a history of neurological diseases or traumatic brain injury
4. Participant has recent suicide attempt leading to current hospital admission or continued expressed suicidal ideation
5. Subject has significant current suicidal ideation within 30 days prior to Screening as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) completed at Screening, that, in the opinion of the investigator, warrants exclusion from the trial
6. Females who are pregnant or lactating
7. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Participants between 18 and 50 years of age with a history of dependence on prescription or non-prescription opioids
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Short Opioid Withdrawal Scale Gossop (SOWS-Gossop) | Daily throughout the 14-day inpatient detoxification treatment
  Correlation of opioid withdrawal symptoms, as measured by the SOWS-Gossop, over time with biomarkers using the EmbracePlus Smartwatch and Corti Wearable.
Clinical Opioid Withdrawal Scale (COWS) | Daily throughout the 14-day inpatient detoxification treatment
  Correlation of opioid withdrawal symptoms, as measured by the COWS, over time with biomarkers using the EmbracePlus Smartwatch and Corti Wearable.
Opioid Craving Visual Analog Scale (OC-VAS) | Daily throughout the 14-day inpatient detoxification treatment
  Correlation of the intensity of opioid cravings, as measured by the OC-VAS, over time with biomarkers using the EmbracePlus Smartwatch and Corti Wearable.
Adverse Events | Daily throughout the 14-day inpatient detoxification treatment
  The primary safety endpoint will be the proportion of participants who experience one or more adverse events.

OTHER OUTCOMES:
Sleep Duration | Daily throughout the 14-day inpatient detoxification treatment
  Correlation of sleep duration and quality with opioid withdrawal symptoms as well as cravings
Stress Monitoring and Assessment Tool (SMART) | Daily throughout the 14-day inpatient detoxification treatment
  Correlation of stress score, as measured by the SMART, with biomarkers using the EmbracePlus Smartwatch and Corti Wearable.
Therapy Compliance | Daily throughout the 14-day inpatient detoxification treatment
  Correlation of compliance to recovery-related therapies (e.g. group therapy, individual counseling) with biomarkers using the EmbracePlus Smartwatch and Corti Wearable.
Drug Screening | Once daily on screening/baseline day, study day 7, and study day 14 (14-day time frame)
  Proportion of participants testing positive for Amphetamines, Buprenorphine, Benzodiazepines, Cocaine, Ethyl Glucuronide, Fentanyl, Synthetic Marijuana, Ecstasy, Methamphetamines, Methadone, Opiates / Morphine, Oxycodone, Cannabinoid (Marijuana), Xylazine, and Tramadol or any combination
Medication Use | Daily throughout the 14-day inpatient detoxification treatment
  Medication use and timing (medication name, dosage, and indication)
Wearable Sensors Compliance | Daily throughout the 14-day inpatient detoxification treatment
  Compliance to wearing wearable sensors (EmbracePlus Smartwatch and Corti Sensor)

CONTACTS AND LOCATIONS:
Overall Officials: Navid Khodaparast, PhD, Principal Investigator — Chief Science Officer; Melanie McWade, PhD, Study Director — Senior Director of Clinical Operations; Carlos Tirado, MD, Study Chair — Medical Monitor
Locations (2):
- United States (2):
  - Hazelden Betty Ford Foundation, Center City, Minnesota
  - Battelle Memorial Institute, Columbus, Ohio

DOCUMENTS (1):
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT06487533/ICF_001.pdf